CLINICAL TRIAL: NCT05930158
Title: The Effectiveness of Dual-task Exercises in Individuals With Chronic Obstructive Pulmonary Disease
Brief Title: The Effectiveness of Dual-task Exercises in Individuals With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, begumunlu, Msc, PT, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 136
Record Dates: First submitted 2023-06-14; First posted 2023-07-05 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: COPD; Healthy
Keywords: COPD; dual-task; balance; walking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pulmonary Rehabilitation Group (Active Comparator): Patients in this group will continue the classic rehabilitation programs determined in the Pulmonary Rehabilitation Unit. The program will continue for 8 weeks, 2 sessions per week.
  Interventions: Other: Pulmonary Rehabilitation
- Dual Task Exercises Group (Experimental): The patients in this group will continue the determined rehabilitation programs, during the walking and balance exercises in the program, they will also do the cognitive exercises that are different from the patients in the Pulmonary Rehabilitation group. The program will continue for 8 weeks, 2 sessions per week. Walking exercises and balance exercises will be planned for 15 minutes each. The intensity of the walking exercise will be planned as moderate intensity according to the results of 6 MWT, it will start with the warm-up period and end with a cool-down. A treadmill will be used for the exercise.
  Balance exercises program will consist of tandem walking (walking with the heel touching the toe of the other foot), standing on one foot (eyes open-closed), walking in a straight line, and standing on soft ground with eyes closed.
  Cognitive exercises to be added during walking and balance exercises will be given as a dual task.
  Interventions: Other: Dual Task Exercises; Other: Pulmonary Rehabilitation
- Healthy Controls (No Intervention): Dual-task performances of healthy individuals with similar demographic characteristics in COPD patients will be compared. For this, the demographic information of healthy volunteers will be recorded, and the Timed Up and Go Test, which will be done as a dual task and a single task, and the 10-meter Walk Test will be evaluated.

INTERVENTIONS:
Other: Dual Task Exercises — Cognitive exercises to be added during walking and balance exercises will be given as a dual task. Cognitive exercises will consist of exercises for memory, executive functions, calculation, information processing speed (reaction time) and working memory areas. Cognitive exercises such as grouping the words given, giving appropriate answers to the simple situations described, simple addition, subtraction, multiplication, and asking the words that the patient is asked to remember before the exercise will be used. Cognitive exercises will be performed simultaneously with walking and balance exercises.
  Arms: Dual Task Exercises Group
Other: Pulmonary Rehabilitation — Pulmonary Rehabilitation content; relaxation exercises, stretching exercises, strengthening exercises, walking exercises, cycling exercises, balance exercises. Exercise intensity will be planned as moderate intensity. Walking and cycling exercises will have warm-up and cool-down periods.
  Arms: Dual Task Exercises Group; Pulmonary Rehabilitation Group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of dual-task performance on motor and cognitive functions and to determine the effect of dual-task exercises given together with the pulmonary rehabilitation program on cardiopulmonary and musculoskeletal parameters in COPD.

The main question[s]it aims to answer are:

* Is dual-task performance in individuals with COPD different from healthy individuals?
* Are dual-task exercises affect cardiopulmonary and musculoskeletal parameters in individuals with COPD? Patients will be randomly divided into 2 groups (Pulmonary Rehabilitation Group, Dual Task Exercises Group). 8-week exercise program will include pulmonary rehabilitation and dual-task exercise group will do their walking and cycling exercises as dual task with another cognitive exercise.

Researchers also will compare (Pulmonary Rehabilitation Group, Dual Task Exercises Group) to see if there is a difference in cardiopulmonary and musculoskeletal parameters.

Researchers also will compare [COPD patients and Healthy Controls] to see if there is a difference in dual-task performance.

DETAILED DESCRIPTION:
Central nervous system dysfunction is an extrapulmonary complication of chronic obstructive pulmonary disease (COPD). Brain functions, particularly frontal lobe functions, have been shown to be impaired as a result of COPD. Studies have shown that patients with COPD have impaired ability to perform complex multitasking, such as driving or walking, along with a cognitive task. It has also been reported that the time to complete a functional test with a cognitive task is prolonged in patients with COPD. For many activities of daily life, it is very important to perform multiple tasks at the same time (such as maintaining balance with a cognitive task) in patients with COPD. Studies evaluating dual-task performance in COPD patients are limited. Since this is an important clinical issue, the reversibility of this situation should also be investigated. In addition, considering the positive effects of pulmonary rehabilitation on cognitive functions such as planning, selective attention and verbal memory, additional dual-task exercises may be an appropriate treatment method and increase the effectiveness of pulmonary rehabilitation and the quality of life of patients.

The aim of this study is to evaluate the effect of dual-task performance on motor and cognitive functions in COPD and to determine the effect of dual-task exercises given together with the pulmonary rehabilitation program on cardiopulmonary and musculoskeletal parameters.

The research will be carried out at the University of Health Sciences Süreyyapaşa Chest Diseases and Thoracic Surgery Training and Research Hospital between June 2023 and November 2024. Patients with a diagnosis of COPD who were admitted to Pulmonary Rehabilitation, met the inclusion criteria, and voluntarily agreed to participate in the study will be included. Demographic information (age, occupation, height, body weight, etc.), clinical status (duration of diagnosis, disease severity), medical conditions, exacerbations and hospitalizations of all participants will be recorded. COPD Assessment Test (CAT) will be administered, and dyspnea evaluation will be made with the Modified Medical Research Council Dyspnea Scale (mMRC). Mini-Mental State Examination and Frontal Assessment Battery will be used in the cognitive status evaluation of the patients. For balance evaluation, it will be done with Mini-BESTest: Balance Evaluation Systems Test. Functional balance and mobility assessment will be made with the Timed Up and Go Test and the 10-meter Walk Test, and the tests will be applied twice as both a single task (normal walking) and a dual task (walking and cognitive task). 6 Minute Walk Test will be used in functional capacity evaluation. Quality of life will be assessed with St. George's Respiratory Questionnaire (SGRQ). In addition, the results of the Pulmonary Function Test performed during the routine controls of the patients will be taken. Patients will be randomly divided into 2 groups (Pulmonary Rehabilitation Group, Dual Task Exercises Group). Evaluations will be repeated at the end of the 8-week exercise program.

Dual-task performances of healthy individuals with similar demographic characteristics in COPD patients will be compared. For this, the demographic information of healthy volunteers will be recorded, and the Timed Up and Go Test, which will be done as a dual task and a single task, and the 10-meter Walk Test will be evaluated.

SPSS (Statistical Package for Social Sciences) (SPSS Inc, IBM Corp, Armonk, New York) statistical program will be used in the classification of the data to be obtained in the research, using qualitative and quantitative statistical methods. With the values in the 95% confidence interval, the significance will be evaluated at the p<0.05 level. In the examination of the variables, appropriate statistical tests will be applied depending on the provision of the parametric test conditions.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with COPD
* COPD patients aged 40-75 years
* COPD stable period
* Absence of abnormal laboratory findings
* Not having a mental problem that prevents them from completing the questionnaires to be - used in the research
* No diagnosed cardiac or pulmonary disease for the healthy control group

Exclusion Criteria:

* COPD exacerbation
* Cognitive impairment
* Having a pregnancy status
* Having advanced age
* Having ischemic heart disease
* Kyphoscoliosis, advanced postural disorder
* Having an orthopedic disability and amputation surgery
* Presence of any neurological disease that causes balance problems
* Having a different respiratory disease that impairs respiratory functions
* Pulmonary embolism
* Pleural effusion
* Heart failure

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Change in Mini-Mental State Exam Score | Baseline and the end of the 8 weeks exercise program
  Mini-Mental State Exam will be used for cognitive status assessment. Mini-Mental State Exam is evaluated out of a total score of 30. Traditionally, scores between 24 and 30 are considered normal. A score below 24 indicates cognitive impairment. The assessment can be completed in 10 minutes. Change from baseline at the end of 8 weeks exercise program will be assessed. Healthy Controls' assessment will be only at the baseline.
Change in Frontal Assessment Battery Score | Baseline and the end of the 8 weeks exercise program
  The Frontal Assessment Battery will be used for cognitive status assessment. It has 6 items and each item has a score of 0-3. A higher score means better performance. The assessment can be completed in 15 minutes. Change from baseline at the end of 8 weeks exercise program will be assessed. Healthy Controls' assessment will be only at the baseline.
Change in dual-task performance with Timed Up and Go Test | Baseline and the end of the 8 weeks exercise program
  Dual-task Assessment will be done with Timed Up and Go Test. While TUG is being performed, the participant initially sits on the chair, gets up from the chair with the start command 3 m. He goes to the marked place ahead, returns, and sits down on the chair again. Patients will be given cognitive tasks during the walking test, while the elapsed time is recorded. The assessment can be completed in 10 minutes. Change from baseline at the end of 8 weeks exercise program will be assessed. Healthy Controls' assessment will be only at the baseline.
Change in dual-task performance with 10 meter Walk Test | Baseline and the end of the 8 weeks exercise program
  Dual-task Assessment will be done with Timed Up and Go Test and 10 meter Walk Test. For 10-meter Walk Test participants are asked to walk 14m during the test. The first 2 m section of the walkway to be applied is the acceleration section, and the last 2 m section is the deceleration section. Patients will be given cognitive tasks during walking test, while the elapsed time is recorded. The assessment can be completed in 10 minutes. Change from baseline at the end of 8 weeks exercise program will be assessed. Healthy Controls' assessment will be only at the baseline.

SECONDARY OUTCOMES:
Change in COPD Assessment Test | Baseline and the end of the 8 weeks exercise program
  CAT is an 8-item unidimensional health status assessment in COPD. Its scoring ranges from 0-40. A higher score denotes a more severe impact of COPD on a person's life. Change from baseline at the end of 8 weeks exercise program will be assessed. The assessment can be completed in 5 minutes.
Change in Dyspnea | Baseline and the end of the 8 weeks exercise program
  Modified Medical Research Council (MMRC) Dyspnea Scale will be used.The patient expresses the degree of dyspnea according to a score between 0-4. The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing. Change from baseline at the end of 8 weeks exercise program will be assessed. The assessment can be completed in 2 minutes.
Change in Balance | Baseline and the end of the 8 weeks exercise program
  Mini-BESTest: Balance Evaluation Systems Test will be used for assessment. It consists of 4 sub-parameters and a total of 14 items. It is a test that is evaluated over a total of 28 points and requires an average of 10-15 minutes. Change from baseline at the end of 8 weeks exercise program will be assessed.
Change in Timed Up and Go Test | Baseline and the end of the 8 weeks exercise program
  Timed Up and Go Test (TUG) will be used to assess functional balance and mobility. While TUG is being performed, the participant initially sits on the chair, gets up from the chair with the start command 3 m. He goes to the marked place ahead and comes back, sits down on the chair again, while the elapsed time is recorded. Change from baseline at the end of 8 weeks exercise program will be assessed. The assessment can be completed in 10 minutes.
Change in 10-meter Walk | Baseline and the end of the 8 weeks exercise program
  10-meter Walk Test will be used for the assessment of functional balance and mobility. For 10-meter Walk Test participants are asked to walk 14m during the test. The first 2 m section of the walkway to be applied is the acceleration section, and the last 2 m section is the deceleration section. Change from baseline at the end of 8 weeks exercise program will be assessed. The assessment can be completed in 10 minutes.
Change in Functional Capacity | Baseline and the end of the 8 weeks exercise program
  6 Minute Walk Test (6MWT) will be used for functional capacity assessment. 6MWT is a test that measures functional exercise capacity, has high structural validity, and shows a high correlation with exercise performance and physical activity scales. The primary endpoint of the test was the six-minute walking distance (6MWM), which is the total distance the patient walked for six minutes. Change from baseline at the end of 8 weeks exercise program will be assessed. The assessment can be completed in 20 minutes.
Change in Quality of Life | Baseline and the end of the 8 weeks exercise program
  Among the tests that measure health-related quality of life, especially St. George's Respiratory Questionnaire (SGRQ) is a test specific for respiratory diseases. SGRQ questions 50 items divided into three areas. Lower scores indicate better health. Change from baseline at the end of 8 weeks exercise program will be assessed. The assessment can be completed in 20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Yıldız Özer, PhD, Study Director — Marmara University
Locations (1):
- University of Health Sciences Süreyyapaşa Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Unlu B, Yildiz Ozer A, Ozmen I, Polat MG. The effectiveness of dual-task exercises in individuals with chronic obstructive pulmonary disease: a study protocol for a randomized controlled trial. Trials. 2025 May 19;26(1):164. doi: 10.1186/s13063-025-08854-2. PMID 40390096